CLINICAL TRIAL: NCT01518712
Title: A Single-Dose, Open-Label, Randomized, 2-Way Crossover Pivotal Study to Assess the Bioequivalence of 2 Fixed Dose Combination Tablets of Canagliflozin and Metformin Immediate Release (IR) (150 mg/850 mg) With Respect to the Individual Components of Canagl
Brief Title: A Study to Assess the Bioequivalence of 2 Fixed Dose Combination (FDC) Tablets of Canagliflozin and Metformin Immediate Release (IR) (150 mg/850 mg) With Respect to the Individual Components of Canagliflozin (1 x 300 mg) and Metformin IR Tablets (2 x 850 mg) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100681; 28431754DIA1052 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2011-12-23; First posted 2012-01-26 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Bioequivalence; Canagliflozin (JNJ-28431754); Metformin IR
MeSH Terms: interventions — Canagliflozin

ARMS (2):
- Treatment Sequence AB (Experimental)
  Interventions: Drug: A (canagliflozin and metformin IR individual tablets) / B (canagliflozin/metformin IR FDC tablets)
- Treatment Sequence BA (Experimental)
  Interventions: Drug: B (canagliflozin/metformin IR FDC tablets / A (canagliflozin and metformin IR individual tablets)

INTERVENTIONS:
Drug: A (canagliflozin and metformin IR individual tablets) / B (canagliflozin/metformin IR FDC tablets) — Treatment A: Canagliflozin: Type = 1, unit = mg, number = 300, form = tablet, route = oral use + metformin IR: Type = 2, unit = mg, number = 850, form = tablet, route = oral use. One canagliflozin tablet and 2 metformin IR tablets taken orally (by mouth) on Day 1 of Treatment Period 1 followed 10-15 days later by Treatment B (canagliflozin/metformin IR FDC): Type = 2, unit = mg, number = 150/850, form = tablet, route = oral use. Two canagliflozin/metformin IR FDC tablets taken orally on Day 1 of Treatment Period 2
  Arms: Treatment Sequence AB
Drug: B (canagliflozin/metformin IR FDC tablets / A (canagliflozin and metformin IR individual tablets) — Treatment B (canagliflozin/metformin IR FDC): Type = 2, unit = mg, number = 150/850, form = tablet, route = oral use. Two Canagliflozin/metformin IR FDC tablets taken orally on Day 1 of Treatment Period 1 followed 10-15 days later by Treatment A: Canagliflozin: Type = 1, unit = mg, number = 300, form = tablet, route = oral use + Metformin IR: Type = 2, unit = mg, number = 850, form = tablet, route = oral use. One canagliflozin tablet and 2 metformin IR tablets taken orally (by mouth) on Day 1 of Treatment Period 2.
  Arms: Treatment Sequence BA

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of fixed dose combination (FDC) tablets of canagliflozin and metformin immediate release (IR) in comparison with the individual components of canagliflozin and metformin IR.

DETAILED DESCRIPTION:
This is an open-label (identity of study drug will be known to volunteer and study staff), single-center study to evaluate the bioequivalence of canagliflozin and metformin IR when administered orally (by mouth) as individual components (ie, separate tablets of canagliflozin and metformin IR) (Treatment A) and when administered as fixed-dose combination (FDC) tablets (ie, canagliflozin and metformin IR contained in the same tablet) (Treatment B). Healthy volunteers participating in the study will be randomly (by chance) assigned to receive Treatment A followed by Treatment B or Treatment B followed by Treatment A with a period of approximately 15 days between treatments.

ELIGIBILITY:
Inclusion Criteria: - Body mass index (BMI) between 18.5 and 30 kg/m² (inclusive) and a body weight of not less than 50 kg. Exclusion Criteria: - History of or current medical illness, abnormal values for hematology or clinical chemistry laboratory tests, or abnormal physical examination, vital signs or 12-lead electrocardiogram (ECG) deemed to be clinically significant by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Canagliflozin plasma concentrations | At 15 time points up to 72 hours
Metformin plasma concentrations | At 13 time points up to 24 hours

SECONDARY OUTCOMES:
Adverse events | Up to approxmately 23 days
  The number and type of adverse events will be reported from Day 1 of treatment period 1 through 7-10 days after treatment period 2 including the 10-15 washout period between treatment periods (total time is approximately 23 days).
Clinical laboratory tests | Up to approxmately 23 days
  Clinically relevant changes occurring in laboratory safety parameters
Vital signs | Up to approximately 23 days
  Blood pressure, pulse, and oral body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Tempe, Arizona, United States